CLINICAL TRIAL: NCT04450719
Title: Exercise Capacity, Muscle Strength, Respiratory Characteristics, Physical Activity and Quality of Life in Patients With Lung Cancer Awaiting Surgery
Brief Title: Pulmonary and Extrapulmonary Impairments in Patients With Lung Cancer Awaiting Surgery
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Professor, Gazi University
Other Study IDs: Gazi University 20
Record Dates: First submitted 2020-06-01; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; walk test; pulmonary functions; muscle strength; physical activity; quality of life
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with lung cancer: Exercise capacity [6-minute walk test (6-MWT)], pulmonary functions [spirometry], respiratory [maximal inspiratory and expiratory pressures (MIP-MEP), mouth pressure device] and peripheral muscle strength [dynamometer], physical activity level [metabolic holter], dyspnea [Modified Medical Research Council dyspnea scale (MMRC)] and quality of life [European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQOL)] were evaluated in patients with lung cancer. Vital signs, dyspnea and fatigue perception [Modified Borg Scale] were recorded as pre-post measurements of 6-MWT.
- Group 2: Healthy individuals: Healthy individuals were selected from individuals without known and diagnosed any chronic diseases. Similar measurements were performed in healthy individuals.

SUMMARY:
To detect comparatively the extent to which physical impairments are observed in patients with lung cancer awaiting lung surgery, comparing exercise capacity, pulmonary functions, muscle strength, physical activity, dyspnea, fatigue and quality of life between the patients with lung cancer and healthy individuals was aimed in current study.

DETAILED DESCRIPTION:
According to global cancer statistics, the most commonly diagnosing and the highest mortality rates belong to lung cancer. As known, patients with lung cancer suffer from many pathophysiological changes due to characteristics of the lung cancer and its cytotoxic treatments including chemotherapy and radiotherapy. Especially, these changes commonly occur in respiratory mechanics and gas exchange all of which resulted in pulmonary function impairment. Moreover, excessive weight loss, anemia, protein catabolism, muscle wasting, skeletal muscle atrophy and inhibition of muscle regeneration are observed in these patients in course of time.

The 6-minute walk test provides valuable and valid knowledge about exercise intolerance in diseases. As known, progressive decline in exercise capacity is commonly observed in patients with lung cancer. The loss of muscle mass also happens not only peripheral muscle but also respiratory muscles in patients with lung cancer. Based on the limited studies regarding patients with lung cancer, weakness in respiratory muscles before surgery has been demonstrated. Furthermore, these patients experience fatigue and dyspnea perceptions all of which increase disease burden and afflict quality of life.

According to the results of a study compared the patients with lung cancer before surgery and healthy individuals, the patients are less physically active than healthy individuals. Moreover, at the diagnosis stage, the patients have worse quadriceps muscle strength, nutritional status, mood and quality of life compared to others. After six months, the patients experience decreases in physical activity, 6-minute walk test distance, and muscle strength and worsening symptoms following chemotherapy, radiotherapy and/or surgery. On the other hand, it could not be clearly demonstrated in the literature to the amount of impairments of pulmonary function and respiratory muscle strength compared to healthy individuals.

To reveal aforementioned impairments in patients with lung cancer before surgery is of importance in terms of being helpful in both determining the protective rehabilitation program and also reducing the disease burden and other possible factors in lung cancer. Therefore, the aim of the current study was to investigate the differences in exercise capacity, pulmonary functions, respiratory and peripheral muscle strength, physical activity level, dyspnea, fatigue and quality of life between the patients with lung cancer before lung surgery and gender and age-matched healthy individuals.

ELIGIBILITY:
Inclusion Criteria for patients:

* being between ages of 18 and 80,
* being a candidate for lung surgery due to lung cancer diagnosis,
* being able to walk,
* receiving optimal medical therapy.

Exclusion Criteria for patients:

* having health problems such as cooperation,
* having orthopedic or neurological disease that limit the walking ability and physical activity,
* having comorbidities such as uncontrolled diabetes mellitus, heart failure, atrial fibrillation and/or hypertension, acute infections,
* having myocardial infarction in the last six months.

Inclusion Criteria for healthy individuals:

* being 18-80 years of age,
* willing to participate to the study,
* being individuals without known and diagnosed any chronic diseases.

Exclusion Criteria for healthy individuals:

* being current smokers,
* being ex-smokers (≥10 pack*years).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty six patients with lung cancer and 21 healthy individuals were included in this study. All patients were referred from Gazi University, Faculty of Medicine, Department of Thoracic Surgery to Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. The patients with lung cancer who were decided to undergo lung surgery by thoracic surgeons were referred to the physiotherapist. Healthy volunteers were also recruited. Then, the patients were matched with healthy individuals according to statistically similarity of both age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6-MWT) | 10 minutes
  Exercise capacity was evaluated with this test according to the guidelines.

SECONDARY OUTCOMES:
Pulmonary function test | 5 minutes
  Dynamic lung volume was measured using a spirometry. Obtained values were represented in percentages.
Respiratory strength test | 10 minutes
  Respiratory muscle weakness was detected using volitional measurements of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) via a portable mouth pressure device based on guidelines. Both MIP and MEP were represented with same units as cmH2O and percentages.
Physical activity measurement | 3 days
  For this evaluation, a metabolic holter was used.
Dyspnea scale | 1 minute
  The Modified Medical Research Council (MMRC) dyspnea scale was used. Dyspnea levels are categorized between 0 (dyspnea only with strenuous exercise) and 4 (too breathless to leave the house or when dressing/undressing).
Quality of life scale | 2 minutes
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version3.0 (EORTC QLQ-C30) was used to evaluate aspects of quality of life impairment. Self-administered questionnaire incorporates five functional scales including social functioning subscale, three symptom scales including fatigue subscale, a global health status and several single items. All item scores are transformed to 0-100. Higher values represent higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased presence of symptoms in symptom scales.
Peripheral muscle strength test | The test was performed during 10 minutes for each participant.
  A hand-held dynamometer was used to evaluate m. quadriceps femoris strength.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — İzmir Democracy University; Ece Baytok, MsC, Study Chair — Gazi University; Zeliha Çelik, MsC, Study Chair — Gazi University; Merve Şatır Türk, MD, Study Chair — Gazi University; Ali Çelik, Prof. Dr., Study Chair — Gazi University; İsmail Cüneyt Kurul, Prof. Dr., Study Chair — Gazi University; Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University Faculty of Health Science Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Jones LW, Eves ND, Haykowsky M, Freedland SJ, Mackey JR. Exercise intolerance in cancer and the role of exercise therapy to reverse dysfunction. Lancet Oncol. 2009 Jun;10(6):598-605. doi: 10.1016/S1470-2045(09)70031-2. PMID 19482248
- [Result] Travers J, Dudgeon DJ, Amjadi K, McBride I, Dillon K, Laveneziana P, Ofir D, Webb KA, O'Donnell DE. Mechanisms of exertional dyspnea in patients with cancer. J Appl Physiol (1985). 2008 Jan;104(1):57-66. doi: 10.1152/japplphysiol.00653.2007. Epub 2007 Nov 1. PMID 17975124
- [Result] Cavalheri V, Jenkins S, Cecins N, Gain K, Phillips M, Sanders LH, Hill K. Impairments after curative intent treatment for non-small cell lung cancer: a comparison with age and gender-matched healthy controls. Respir Med. 2015 Oct;109(10):1332-9. doi: 10.1016/j.rmed.2015.08.015. Epub 2015 Aug 29. PMID 26342839
- [Result] Pinson P, Klastersky J. The value of lung function measurements for the assessment of chemotherapy in lung cancer patients. Lung Cancer. 1998 Mar;19(3):179-84. doi: 10.1016/s0169-5002(97)00094-9. PMID 9631365
- [Result] Granger CL, McDonald CF, Irving L, Clark RA, Gough K, Murnane A, Mileshkin L, Krishnasamy M, Denehy L. Low physical activity levels and functional decline in individuals with lung cancer. Lung Cancer. 2014 Feb;83(2):292-9. doi: 10.1016/j.lungcan.2013.11.014. Epub 2013 Nov 26. PMID 24360323
- [Result] Sullivan MJ, Green HJ, Cobb FR. Altered skeletal muscle metabolic response to exercise in chronic heart failure. Relation to skeletal muscle aerobic enzyme activity. Circulation. 1991 Oct;84(4):1597-607. doi: 10.1161/01.cir.84.4.1597. PMID 1914100
- [Result] Wagner PD. The major limitation to exercise performance in COPD is inadequate energy supply to the respiratory and locomotor muscles vs. lower limb muscle dysfunction vs. dynamic hyperinflation. The real cause of exercise limitation in COPD. J Appl Physiol (1985). 2008 Aug;105(2):758. doi: 10.1152/japplphysiol.90336.2008c. No abstract available. PMID 18678625
- [Result] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613
- [Result] Granger CL, Holland AE, Gordon IR, Denehy L. Minimal important difference of the 6-minute walk distance in lung cancer. Chron Respir Dis. 2015 May;12(2):146-54. doi: 10.1177/1479972315575715. Epub 2015 Mar 6. PMID 25749346
- [Result] Laude EA, Duffy NC, Baveystock C, Dougill B, Campbell MJ, Lawson R, Jones PW, Calverley PM. The effect of helium and oxygen on exercise performance in chronic obstructive pulmonary disease: a randomized crossover trial. Am J Respir Crit Care Med. 2006 Apr 15;173(8):865-70. doi: 10.1164/rccm.200506-925OC. Epub 2006 Jan 26. PMID 16439720
- [Result] Nomori H, Horio H, Fuyuno G, Kobayashi R, Yashima H. Respiratory muscle strength after lung resection with special reference to age and procedures of thoracotomy. Eur J Cardiothorac Surg. 1996;10(5):352-8. doi: 10.1016/s1010-7940(96)80094-7. PMID 8737692
- [Result] Weiner P, Man A, Weiner M, Rabner M, Waizman J, Magadle R, Zamir D, Greiff Y. The effect of incentive spirometry and inspiratory muscle training on pulmonary function after lung resection. J Thorac Cardiovasc Surg. 1997 Mar;113(3):552-7. doi: 10.1016/S0022-5223(97)70370-2. PMID 9081102
- [Result] Bower JE. Cancer-related fatigue--mechanisms, risk factors, and treatments. Nat Rev Clin Oncol. 2014 Oct;11(10):597-609. doi: 10.1038/nrclinonc.2014.127. Epub 2014 Aug 12. PMID 25113839
- [Result] Fox SW, Lyon DE. Symptom clusters and quality of life in survivors of lung cancer. Oncol Nurs Forum. 2006 Sep 1;33(5):931-6. doi: 10.1188/06.ONF.931-936. PMID 16955121